CLINICAL TRIAL: NCT03672409
Title: Diabetes Training Program for Doctors, Nurses and Nutritionists in Primary Health Care in Hermosillo, Sonora
Brief Title: Diabetes Training Program for Health Professionals From Hermosillo, Sonora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Centroid
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Knowledge
Keywords: Knowledge in Type 2 diabetes,; Training program; Primary health care
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention in knowledge (Other): All participants will be offered learning sessions to improve knowledge in diabetes
  Interventions: Behavioral: Intervention in knowledge

INTERVENTIONS:
Behavioral: Intervention in knowledge — The knowledge intervention will be done through four group learning sessions with the objective of significantly increasing diabetes knowledge in health professionals.
  The learning sessions will be carried out weekly in a period of 4 weeks, with a duration of 60 minutes per session. In addition, two sessions will be held for the evaluation of pre and post intervention knowledge. The learning sessions consist in the diagnosis, evaluation, complications and comorbidities, pharmacological treatment and nutrition in type 2 diabetes.
  Other Names: Training program

SUMMARY:
Primary health care is the medical assistance available to all individuals in a community and is considered the core of the health system. Diabetes, among other chronic diseases, is a common reason for medical consultation in primary health care. Worldwide and in Mexico, the prevalence of diabetes has been increasing in recent decades, which also leads to an increase in the number of deaths. On the other hand, the annual cost of medical care for diabetes in the country has increased due to the exacerbation of complications and comorbidities associated, which are presented, among other causes, by a deficiency of knowledge in the diagnosis, evaluation, management and follow-up of type 2 diabetes, of health professionals (doctors, nurses, nutritionists) working in primary health care.

The present study will allow evaluating the effect of a training program, is a single-cohort clinical study with pre- and post-intervention measurements lasting 6 weeks, including the initial and final measurements of health professionals currently working in primary health care of Hermosillo Sonora.

DETAILED DESCRIPTION:
The study aims to improve knowledge in diabetes through the design and evaluation of a training program in health professionals (doctors, nurses and nutritionists) in primary health care.

The hypothesis of the study is that the training program in diabetes aimed doctors, nurses and nutritionists in primary health care will significantly increase knowledge in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, nurses and nutritionists of primary health care in Hermosillo, Sonora.
* Belonging to the health jurisdiction and the general hospital of the state
* That provide consultation to patients with diabetes
* Age 20 years and less than 65
* Desire of participate
* Sign up the consent form

Exclusion Criteria:

* Do not meet the inclusion criteria

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge measurements in diabetes by questionnaire | 6 weeks
  Diabetes training program focused on improving knowledge in primary health care professionals

CONTACTS AND LOCATIONS:
Overall Officials: Julian G Esparza Romero, PhD, Principal Investigator — Centro de Investigación en Alimentación y Desarrollo A.C.
Locations (1):
- Centro de Investigación en Alimentación y Desarrollo, Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Undecided